CLINICAL TRIAL: NCT06616883
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Cross-over Study to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Single Administration of DA-5221_01 and Concomitant Administration of DA-5221_01-R1 and DA-5221_01-R2 Under Fasting Conditions in Healthy Adult Volunteers
Brief Title: Pharmacokinetics and Safety Profiles After Administration of DA-5221_01 and Co-administration of 5221_01-R1 and DA-5221_01-R2 in Healthy Adult Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA5221_01_BE_I
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Sequence A (Experimental)
  Interventions: Drug: DA-5221_01; Drug: DA-5221_01-R1 + DA-5221_01-R2
- Experimental: Sequence B (Experimental)
  Interventions: Drug: DA-5221_01; Drug: DA-5221_01-R1 + DA-5221_01-R2

INTERVENTIONS:
Drug: DA-5221_01 — single dose administration (DA-5221_01 one tablet once a day)
Drug: DA-5221_01-R1 + DA-5221_01-R2 — single dose administration (DA-5221_01-R1 one tablet once a day + DA-5221_01-R2 one tablet once a day)

SUMMARY:
Pharmacokinetics and Safety Profiles After Administration of DA-5221_01 and Co-administration of 5221_01-R1 and DA-5221_01-R2 in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI between 18 and 30 kg/m2
* Body weight: Male≥50kg, Female≥45kg
* Subjects who have signed an informed consent themselves after receiving detailed explanation about clinical study

Exclusion Criteria:

* Subjects with clinically significant medical history
* Subjects with history of drug abuse or addicted

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-18 (Estimated)

PRIMARY OUTCOMES:
AUCt | pre-dose~72 hours post-dose
  area under the curve
Cmax | pre-dose~72 hours post-do
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin Hospital, Seoul, South Korea, South Korea